CLINICAL TRIAL: NCT03718871
Title: Expanding HIV Testing Among Uganda Adults Who Utilize Traditional Healers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Mbarara University of Science and Technology (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1803019105; K23MH111409 (NIH)
Record Dates: First submitted 2018-04-21; First posted 2018-10-25 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: HIV/AIDS; Health Behaviors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a mixed methods study where Aims 1 and 2 have both qualitative and quantitative arms. Aim 3 is an unblinded intervention, with a control arm, to be delivered in cluster-randomized fashion (Sept 2019-June 2020). Healers will be treated as clusters and randomized to either intervention or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healer HIV testing intervention (Experimental): We will follow Ugandan National protocols to administer voluntary HIV testing at 9 TH practice locations throughout Mbarara District over a 9 month period.
  Interventions: Behavioral: HIV testing at traditional healer practices
- Healer control arm (No Intervention): Patients will undergo protcolized usual TH care at 8 practices, which include HIV education and a referral to receive VCT through existing resources. Study staff will contact the client at 3 months following enrollment to assess for self-report of VCT.

INTERVENTIONS:
Behavioral: HIV testing at traditional healer practices — HIV 1/2 antigen-antibody POC test (Oraquick©) will be administered to those participants who agree to test. Pre-test counseling will be performed before results are delivered. Clients with positive tests will be provided with detailed contact information for the MUST ISS clinic, and given specific instructions to present to the clinic as soon as possible for confirmatory testing and linkage to care.
  Arms: Healer HIV testing intervention

SUMMARY:
HIV antiretroviral therapy has the potential to dramatically decrease HIV transmission worldwide1; yet, a barrier to ending the AIDS epidemic in low-resource settings is the fact that healthcare is largely provided by traditional or spiritual healers rather than biomedical providers, and there are no strategies in place to identify HIV-infected patients among Traditional Healer patients and link them to HIV care. In order to reach the UNAIDS 90-90-90 benchmarks HIV services must reach marginalized populations in endemic regions, such as in southwestern Uganda. Uganda is one of seven sub-Saharan African (SSA) countries accounting for 90% of all new HIV infections in this region6. HIV prevalence is 7.3%, with ~1.5 million people living with HIV/AIDS and 99,000 new infections in 2014. However, only 50% of sexually active Ugandans have ever tested for HIV8. In the project location of southwestern Uganda, like much of SSA, the majority of Ugandans utilize Traditional Healers (TH), but little is known about Traditional Healer practices or rates of HIV testing (or HIV infection) among their clients. Specific aims of this study are to: 1) identify key socio-structural factors that frame HIV testing behaviors among Ugandan adults who utilize Traditional Healers; 2) investigate acceptability of providing point-of-care HIV testing at Traditional Healer practice locations; and 3) develop and pilot a prospective HIV testing intervention among Traditional Healer patients to promote earlier diagnosis. Results will be used to implement subsequent, large-scale cluster-randomized HIV testing intervention at Traditional Healer practice locations. Findings from the proposed study include formative data on populations that utilize Traditional Healers in an HIV-endemic region of Uganda, and pilot testing of an HIV testing intervention at healer practice locations; these results could be applied towards expanding HIV testing in other low-resource, endemic settings.

DETAILED DESCRIPTION:
This study has three specific aims:

Specific Aim 1: Identify key socio-structural factors that frame HIV testing behaviors among clients of Ugandan TH, using an exploratory sequential, mixed-methods study design. First, qualitative interviews with 25-35 purposely-sampled TH clients will characterize the care-seeking trajectory, HIV testing behaviors and related stigma, healthcare costs, and HIV risks and exposures. Based on these results, a survey will be designed and administered to 300 Ugandan adults who utilize TH in Mbarara District. This cross-sectional study will identify 1) rates of HIV testing among TH clients and 2) variables that independently predict HIV testing within the prior 12 months. These data will inform a model of HIV testing behavior among TH clients based on the Andersen Model of Healthcare Utilization, and generate hypotheses to be tested in Specific Aim 2.

Specific Aim 2: Characterize acceptability of receiving point-of-care (POC) HIV testing at TH locations, using an exploratory sequential, mixed-methods approach. Qualitative interviews with 15-25 purposely sampled TH and 15-25 purposely-sampled TH clients will explore attitudes and experiences with biomedicine, feasibility and acceptability of delivering POC HIV testing at TH locations, and investigate relevant themes emerging from Aim 1. Based on qualitative results, a survey will be developed and administered to 175 TH in Mbarara District. This cross-sectional study will characterize TH practices relevant to HIV testing, and identify characteristics of healers who favorably view the proposed intervention (Specific Aim 3). These data will be integrated with results from SA1 to develop an intervention that will overcome socio-structural barriers to HIV testing.

Specific Aim 3: Develop and pilot an HIV testing intervention among TH clients using a cluster randomized study design. Integration of results from SA1 and SA2 will inform a pilot HIV testing intervention at 9 TH practice locations, to be compared with a control group receiving usual TH care at 8 practices. This pilot will offer HIV testing at TH practice sites to 250 TH clients at the intervention arm sites, and offer protocoled usual care to 250 clients at control arm sites. Primary outcome for this study will be rates of HIV testing among TH clients. Secondary outcomes will include i) number of new HIV diagnoses among TH clients, and ii) number of patients with +HIV POC test who successfully link to HIV care in 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age or older
* able to provide informed consent
* not known to be HIV infected
* willing to be contacted at 3 months following enrollment
* willing to complete an exit survey after 3 months

Exclusion Criteria:

* being under the age of 18 years
* incapable of giving informed consent
* previously being diagnosed with HIV
* being unwilling to receive HIV test results
* unwilling to participate in the testing intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Sundararajan, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
De-identified IPD may be shared with other researchers with reasonable, written requests, and approval from all researchers involved with this current study.

REFERENCES:
- [Derived] Sundararajan R, Ponticiello M, Lee MH, Strathdee SA, Muyindike W, Nansera D, King R, Fitzgerald D, Mwanga-Amumpaire J. Traditional healer-delivered point-of-care HIV testing versus referral to clinical facilities for adults of unknown serostatus in rural Uganda: a mixed-methods, cluster-randomised trial. Lancet Glob Health. 2021 Nov;9(11):e1579-e1588. doi: 10.1016/S2214-109X(21)00366-1. PMID 34678199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 traditional healers practicing within an eight-kilometer distance from Mbarara Township were screened for eligibility.
Pre-assignment Details: Five healers were excluded due to self-reported weekly volume <7 patients. Three healers declined to participate because of scheduling conflicts. On August 2, 2019 the remaining 17 healers were randomized into two study arms (9 to intervention, 8 to control. From August 8, 2019-February 7, 2020, 500 participants were enrolled at healer cluster sites
Units Other Than Participants: Traditional healer practices
Groups:
- Healer Control Arm: Patients will undergo protocolized usual care at 8 healer practices, which includes HIV education and a referral to receive voluntary HIV testing at local medical clinics.
- Healer HIV Testing Intervention: 9 healers will deliver pre-test counseling and offer HIV 1/2 antigen-antibody POC test (Oraquick©) to eligible participants. Post-test counseling will be delivered and those testing positive will be provided information about where to receive linkage to HIV care.
Period: Overall Study
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Started | 250; 8 Traditional healer practices | 250; 9 Traditional healer practices
Completed | 250; 8 Traditional healer practices | 250; 9 Traditional healer practices
Not Completed | 0; 0 Traditional healer practices | 0; 0 Traditional healer practices

BASELINE CHARACTERISTICS:
Groups:
- Healer Control Arm: Patients will undergo protcolized usual care at 8 healer practices, which include HIV education and a referral to receive VCT through local HIV testing clinics. Study staff will contact the client at 3 months following enrollment to assess for self-report of VCT.
- Healer HIV Testing Intervention: HIV testing at traditional healer practices: HIV 1/2 antigen-antibody POC test (Oraquick©) will be administered to those participants who agree to test. Pre-test counseling will be performed before results are delivered.
- Total: Total of all reporting groups
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [24 to 39] | 28.5 [23 to 38] | 29 [24 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 134 | 279
  Male | 105 | 116 | 221
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of participants who completed primary education or lower [Count of Participants; unit: Participants] | 139 | 143 | 282
Number of participants who are Christian [Count of Participants; unit: Participants] | 218 | 237 | 455
Number of participants who are married [Count of Participants; unit: Participants] | 164 | 142 | 306

OUTCOME MEASURES:

1. Primary Outcome: Number of TH Clients Who Received HIV Testing
Description: Primary study outcome was receipt of an HIV test within 90 days of enrollment. In the control arm, this was assessed via self-report at time of 90-day phone call follow up. For intervention arm, the participating healer recorded whether an HIV test was accepted by the participant at the time of the study visit. If the HIV test was accepted and delivered, the healer recorded the result of the test.
Time Frame: within 3 months following study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 250 | 250
Participants | 57 | 250
Statistical Analysis 1: Comparison: Healer Control Arm vs Healer HIV Testing Intervention; Given that the intervention arm showed 100% uptake, a multi-level regression model could not be created with a zero in the denominator in the intervention group. We therefore used Fisher's exact test to assess for significant differences in proportion of HIV testing between study arms; Test type: Superiority; p < 0.001, Fisher Exact — The threshold for significance was set at p < 0.05; intracluster correlation coefficient = 0.086, 95% CI 2-sided [0.015 to 0.363]

2. Secondary Outcome: Number of New HIV Diagnoses Among TH Clients
Description: For intervention arm participants, the healer recorded the result of the point-of-care HIV test for those participants who agreed to test during the study visit. In the control arm, this outcomes was assessed via self-report during the 90-day follow up phone call.
Time Frame: within three months following enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 250 | 250
Participants | 0 | 10
Statistical Analysis 1: Comparison: Healer Control Arm vs Healer HIV Testing Intervention; Test type: Superiority; p = 0.002, Fisher Exact

3. Secondary Outcome: Number of Patients With +HIV Test Who Successfully Link to HIV Care
Description: This outcome was assessed via self-report during the 90-day follow up phone call. For participants newly testing HIV-positive, questions were posed to determine if they had received confirmatory testing, and initiated ART medication.
Time Frame: at three months following enrollment.
Population: Zero participants in the control arm were newly diagnosed with HIV infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 250 | 250
Participants | 0 | 7
Statistical Analysis 1: Comparison: Healer Control Arm vs Healer HIV Testing Intervention; Test type: Superiority; p = 0.015, Fisher Exact

4. Secondary Outcome: Age in Years of Control Arm Subjects Who Received an HIV Test
Description: Participants in the control arm assessed for primary outcomes of receiving an HIV test within 3 months of study enrollment. Participant age in years at time of study enrollment, and association with primary outcome of receiving an HIV test
Time Frame: 3 months following study enrollment
Population: Only control arm participants who received an HIV test were included in this analysis, as all intervention arm participants accepted an HIV test as part of the study and therefore, no other variates would be statistically associated with receiving a test more than being in the intervention study arm.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 57 | 0
years | 30 [24 to 39] |
Statistical Analysis 1: Comparison: Healer Control Arm; We considered variables that predicted the primary outcome of receiving an HIV test among control arm only, as uptake was 100% in the intervention. First we identified variables that were significant (two-sided p-value<0.05) in univariate analysis and creating multivariate mixed-effects logistic regression model accounting for covariates and intercorrelation between participants from the same healer by including healers as random effects; Test type: Other — No comparison between study arm groups was made in this analysis, as it was limited to control arm only; p < 0.01, Regression, Linear — Significance threshold two-sided alpha = 0.05; Odds Ratio (OR) = 1.04, 95% CI 2-sided [1.02 to 1.06], Standard Deviation 0.039

5. Secondary Outcome: Gender of Control Arm Subjects Who Received an HIV Test
Description: Self-reported participant gender and association with primary study outcome of receiving an HIV test
Time Frame: at 3 months following enrollment
Population: Participants in the control arm assessed for primary outcomes of receiving an HIV test within 3 months of study enrollment. Only control arm participants were included in this analysis, as all intervention arm participants accepted an HIV test as part of the study and therefore, no other variates would be statistically associated with receiving a test more than being in the intervention study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 57 | 0
Participants
  Males | 17 |
  Females | 40 |
Statistical Analysis 1: Comparison: Healer Control Arm; [analysis description as in outcome 4, analysis 1]; Test type: Other — No comparison was made with the intervention arm; p = 0.07, Fisher Exact — Univariate analysis; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.30 to 1.04]

6. Secondary Outcome: Highest Level of Education for Control Arm Subjects Who Received an HIV Test
Description: Participant self-reported highest level of education, and association with study primary outcome of receiving an HIV test
Time Frame: at 3 months following study enrollment
Population: We considered variables that predicted the primary outcome of receiving an HIV test among control arm only, as uptake was 100% in the intervention. First we identified variables that were significant (two-sided p-value<0.05) in univariate analysis and creating multivariate mixed-effects logistic regression model accounting for covariates and intercorrelation between participants from the same healer by including healers as random effects.
Measure: Count of Participants; unit: Participants
Groups:
- Healer HIV Testing Intervention: HIV testing at 9 traditional healer practices: HIV 1/2 antigen-antibody POC test (Oraquick©) will be administered to those participants who agree to test. Pre-test counseling will be performed before results are delivered.
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
Number analyzed (Participants) | 57 | 0
Participants
  Primary school education or lower | 30 |
  Secondary school education or higher | 27 |
Statistical Analysis 1: Comparison: Healer Control Arm; [analysis description as in outcome 4, analysis 1]; Test type: Other — Comparison between study arms was not performed; p = 0.09, Fisher Exact; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.16 to 1.18]

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Healer Control Arm | Healer HIV Testing Intervention
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250 | 0/250
Other Adverse Events (participants affected / at risk) | 0/250 | 0/250

LIMITATIONS AND CAVEATS:
Our goal was to evaluate the effectiveness of delivering HIV testing via a novel implementation strategy. This was not a large-scale cost-effectiveness trial. Future studies are needed to evaluate program cost. Since we excluded healers with the lowest patient volume, results may not be generalizable to these smaller practices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT03718871/Prot_SAP_000.pdf